CLINICAL TRIAL: NCT06273475
Title: The Effect of Robot-Assisted Versus Standard Training on Motor Function Following Subacute Rehabilitation After Ischemic Stroke - a Randomised Controlled Trial Nested in a Prospective Cohort.
Brief Title: Robot-Assisted Training Versus Standard Training in Ischemic Stroke
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Odense University Hospital (Other)
Collaborators: University of Southern Denmark (Other); Rigshospitalet, Denmark (Other); Herlev and Gentofte Hospital (Other); Stanford University (Other); Sygehus Lillebaelt (Other); Danish Association of the Physically Disabled (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: OUH RoboRehab
Record Dates: First submitted 2024-02-01; First posted 2024-02-22 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-05

CONDITIONS: Stroke; Ischemic Stroke
Keywords: Stroke; Body weight unloading; Motor function; Rehabilitation
MeSH Terms: conditions — Stroke; Ischemic Stroke

STUDY DESIGN:
Intervention Model Description: Multicentre randomised (1:1) parallel-group intervention study with assessor-blinding.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Data will be analysed by the PhD student blinded towards group allocation. The test leader responsible for RCT outcome assessment will be blinded towards group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Training facilitated through body weight unloading robotic technology yielding a dynamic unloading force applied to the body centre of mass.
  Interventions: Other: Robot-assisted Training
- Active Control (Active Comparator): Training facilitated without the use of body weight unloading robotic technology, thereby only allowing manual assistance from physiotherapists.
  Interventions: Other: Standard Training

INTERVENTIONS:
Other: Robot-assisted Training — Gait training and functional strength training facilitated by body weight unloading robotic technology yielding a dynamic unloading force applied to the body centre of mass. Gait training will be conducted both on treadmill and overground. Functional strength training exercises include sit-to-stand, stair-walking, step-ups etc. The goal is to gradually reduce body weight unloading as participants progress through the intervention period.
  Arms: Intervention
Other: Standard Training — Gait training and functional strength training facilitated without the use of body weight unloading robotic technology, thereby only allowing manual assistance from physiotherapists. The goal of training is the same as in the intervention group, however no body weight unloading device will be implemented in the active control group.
  Arms: Active Control

SUMMARY:
The aim of this randomised controlled trial (RCT) nested in a prospective cohort, is to investigate the superior effect of late-phase robot-assisted versus standard training on motor function, physical function, fatigue, and quality of life in a moderately-to-severely impaired chronic stroke population following subacute rehabilitation.

The main hypothesis of the study is:

Robot-assisted training has a superior effect on motor function (Fugl-Meyer Lower Extremity Assessment; primary outcome), physical function, fatigue, and quality of life in moderately-to-severely impaired chronic stroke-affected individuals in comparison to standard training.

DETAILED DESCRIPTION:
Background:

Stroke is the collective term for acute focal injuries to the central nervous system (CNS) caused by a disturbance in the blood circulation of the brain i.e., cerebral infarction (ischemic stroke) or intracerebral hemorrhage (hemorrhagic stroke). On an annual basis, 113,000 UK citizens and 12,000 Danish citizens are hospitalised following a stroke, and worldwide stroke is one of the leading causes of disability. Stroke-affected individuals may display residual impairments in motor, physical and cognitive functions along with mental fatigue and depression. Body weight unloading (BWU) has been suggested as a method of training for people with neurological disorders suffering from severe limitations in walking ability. BWU is the application of a vertical upwards force on the body centre of mass, thereby alleviating individuals of supporting their own body weight against gravity. However, the efficacy of BWU-based training is unclear. Therefore, the aim of the present study is to investigate the superior effect of late-phase robot-assisted versus standard training on motor function, physical function, fatigue, and quality of life in a moderately-to-severely impaired chronic stroke population following subacute rehabilitation.

Trial design overview:

Randomised, assessor-blinded, two-arm, multicentre trial. Participants will be recruited through Odense University Hospital, Herlev Gentofte Hospital and Rigshospitalet. Stroke-affected patients are recruited to the prospective cohort 3 months post-stroke. Stroke-affected individuals will be recruited to the RCT from the prospective cohort 6 months post-stroke and randomised 1:1 for robot-assisted training (intervention group) or standard training (active control group). Cohort participants not eligible and/or interested in participation in the RCT study will continue their participation in the prospective cohort.

The RCT study compares training with the robot-assisted body weight unloading to standard training without the robot. Training programs will be matched for total hours allocated to training and will consist of 2 sessions per week with a physiotherapist (one-on-one) and last 6 months (48 training sessions in total). Each session will last 60 minutes, 75 minutes and 90 minutes during the first, middle and last two months of the training program, respectively. Thus, INT and CON are matched for training time, but the effective training volume (resistance times repetitions) is not controlled.

Blinding:

The primary investigator will be blinded to allocation and will not participate in the randomisation, training or testing of participants. Statistical analysis will be performed on allocation codes. The test leader responsible for RCT-study testing will be blinded. It will not be possible to blind study participants and the physiotherapists conducting the training.

Randomisation Randomisation is performed internet-based using REDCap Randomise allocated 1:1. The randomisation takes place following pre-intervention testing at 6-months post-stroke. The study uses block randomisation in blocks of 2 and 4. Stratification is applied using the Modified Rankin Scale (3,4,5). The primary investigator is blinded with respect to the permuted blocking strategy. A data manager with no clinical involvement in the trial, prepares the randomisation sequence, and the allocation is concealed in a password-protected computer file.

Compliance

No study restrictions are imposed on potential regular 'outside-the-study' visits to physiotherapist or visits from occupational therapists. Acceptable adherence is defined as a completion of minimum 70% of scheduled sessions. Moreover, number/percent of completed training sessions and achievement of target intensity/volume will be registered in a training log by the physiotherapist.

Time points

Time points are reported as time since onset of stroke. The following time-points are therefore included in the present study: 3-, 6-, 12-, and 18-months post-stroke (corresponding to T3, T6, T12 and T18). Onset of stroke is indicated as T0.

Questionnaires are sent to the prospective cohort participants at T3, T6, T12, T18. RCT-outcomes will be assessed at pre-intervention (T6) and post-intervention (T12). Blood samples will be included at T3, T6, T12.

Sample Size

A priori sample size calculation was performed and resulted in a required sample size of 34 study participants. This was based on detecting a minimally clinically important between-group difference (MCID) of 6 points on the FM-LE scale and a standard deviation of 6 points at an α level of 5% and with a statistical power of 80%. Allowing for dropout the aim is to include 40 participants in total.

Statistical analysis

An assessor-blinded intention-to-treat (ITT) analysis will be performed on primary and secondary outcome measures (Primary Analysis). A full analysis data set will be created with two imputation techniques and sensitivity analysis will be performed to examine robustness of any statistically significant differences. The ITT analysis will employ a two-way analysis of variance (ANOVA) to analyse between-group differences in change-scores from pre- to post-intervention. A per protocol analysis (between-group differences in change-scores using ANOVA) will be included as a secondary analysis on participants demonstrating acceptable adherence (>70%).

Ethics:

The study was submitted to The Regional Committees on Health Research Ethics for Southern Denmark. The project approved the project on the 17th of January 2024.

ELIGIBILITY:
Inclusion:

1. Ischemic and haemorrhagic stroke
2. Chronic state (6-24 months post-stroke).
3. Subacute rehabilitation terminated (subacute phase defined as until 6 months post-stroke).
4. Moderately-severely impaired:

   1. Modified Rankin Scale Score 3-5.
   2. Scandinavian Stroke Scale Leg Motor Function Score 0-4 and/or SSS gait function 0-9.
5. Approved by referring doctor

Exclusion:

1. Prior SAH
2. Infarct located in the cerebellum or brain stem
3. Severe fatigue making study completion improbable.
4. Cognitive deficits impeding study participation.
5. Inability to walk independently pre-stroke.
6. Recurrence of cardiovascular/cerebrovascular accidents.
7. Pre-existing neurological diseases or ongoing cancer treatment.
8. Refusing group allocation.
9. Concurrent participation in another clinical trial potentially interacting with the present trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-05-01 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2027-02-01 (Estimated)

PRIMARY OUTCOMES:
Fugl-Meyer Lower Extremity Assessment of Motor Function | Pre-intervention (6-18 months post-stroke) and post-intervention (12-24 months post-stroke).
  The primary outcome measure is the between-group difference in change score of Fugl-Meyer Lower Extremity Assessment (FM-LE) from pre- (T6) to post-intervention (T12). The FM-LE assesses motor function and has been recommended as a part of a core outcome set in stroke rehabilitation studies.

SECONDARY OUTCOMES:
Modified Rankin Scale Score (between-group change) | Prospective cohorte: 3, 6, 12, and 18 months post stroke. RCT: Pre-intervention (6-18 months post-stroke) and post-intervention (12-24 months post-stroke) and follow-up (18-30 months post-stroke).
  Global disability will be assessed using the Modified Rankin Scale, which classifies participants from 0-6 as 0) no symptoms, 1) no significant disability, 2) slight disability, 3) moderate disability, 4) moderate severe disability, 5) severe disability and 6) deceased.
Functional Ambulation Category (between-group change) | RCT: Pre-intervention (6-18 months post-stroke) and post-intervention (12-24 months post-stroke).
  The Functional Ambulation Category is a clinical gait assessment scale used to distinguish 6 levels of walking ability based on required physical support. The categories are as follows: 0) Nonfunctional ambulation, 1) Ambulator - Dependent for Physical Assistance Level 2, 2) Ambulator - Dependent for Physical Assistance Level 1, 3) Ambulator - Dependent for Supervision, 4) Ambulator - Independent, Level surfaces only, 5) Ambulator - Independent.
Berg Balance Scale (between-group change) | RCT: Pre-intervention (6-18 months post-stroke) and post-intervention (12-24 months post-stroke).
  The Berg Balance Scale consists of 14 items testing the participant's ability to maintain positions of varying difficulty and to perform tasks such as transfer between positions, reach forward and alter stance positions. Each item is scored on a five-point ordinal scale ranging from 0 (cannot perform the task) to 4 (independence). Total scores can range from 0 to 56.
Barthel-100 Index (between-group change) | RCT: Pre-intervention (6-18 months post-stroke) and post-intervention (12-24 months post-stroke).
  The Barthel-100 Index is a clinical assessment of independence in activities of daily living (ADLs) through observation. The assessment has 10 items (feeding, bathing, grooming, dressing, bowels, bladder, toilet use, transfers, mobility, stairs) and participants may score 0-100 points. This measurement has been recommended as a part of a core outcome set.
Global Rating of Change (between-group change) | RCT: Post-intervention (12-24 months post-stroke) and follow-up (18-30 months post-stroke)
  Global Rating of Change is used to assess the participants' overall experience of change from pre- to post-intervention (T6-T12) and from post-intervention to follow-up (T12-T18). A seven-point likert scale is used. Participants will be asked to compare their current overall health to their health 6 months ago with answers ranging from "Much worse", "Little worse", "The same", "Little better", and "Much better.
International Physical Activity Questionnaire - Short Form (between-group change) | Prospective cohorte: 3, 6, 12, and 18 months post stroke. RCT: Pre-intervention (6-18 months post-stroke) and post-intervention (12-24 months post-stroke) and follow-up (18-30 months post-stroke).
  The International Physical Activity Questionnaire - Short Form is a patient-reported outcome measurement used to measure physical activity over the past week in four different intensity levels, including 1) vigorous activities, 2) moderate activities, 3) walking, and 4) sitting. Higher values equal higher levels of physical activity.
Fatigue Severity Scale 7 (between-group change) | Prospective cohorte: 3, 6, 12, and 18 months post stroke. RCT: Pre-intervention (6-18 months post-stroke) and post-intervention (12-24 months post-stroke) and follow-up (18-30 months post-stroke).
  The Fatigue Severity Scale 7 (FSS-7) is a one-dimensional 7-item patient reported outcome measurement commonly implemented in stroke trials. Each item is scored from one to seven with higher scores indicating increased fatigue. The FSS-7 was shown to be more valid than the 9-item version of the instrument (FSS-9), and therefore this version of the instrument is implemented.
EQ-5D-5L Quality of Life (between-group change) | Prospective cohorte: 3, 6, 12, and 18 months post stroke. RCT: Pre-intervention (6-18 months post-stroke) and post-intervention (12-24 months post-stroke) and follow-up (18-30 months post-stroke).
  The EQ-5D-5L (European Quality of Life - 5 Dimensions) is a validated survey for measuring health-related quality of life. It consists of five dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. The outcome is reported on a scale of 1-5 where 1 is no problems and 5 is extreme problems. This measurement has been recommended as a part of a core outcome set.
Hand-grip strength (between-group change) | RCT: Pre-intervention (6-18 months post-stroke) and post-intervention (12-24 months post-stroke).
  Hand-grip strength is a performance-based measurement assessed using a hand-held dynamometer. The outcome is in kilograms and used in the present study as an indicator for upper limb function.
Gait speed (between-group change) | RCT: Pre-intervention (6-18 months post-stroke) and post-intervention (12-24 months post-stroke).
  The 10-meter walking test is a performance-based measurement to evaluate gait speed. This test is recommended in two forms as a part of a core outcome set; 1) Can the person independently walk 10 metres (gait aids permitted) yes/no? and 2) gait speed on the 10-meter test if the person is able to independently walk 10 metres.

OTHER OUTCOMES:
Muscle Strength (between-group change) | RCT: Pre-intervention (6-18 months post-stroke) and post-intervention (12-24 months post-stroke).
  Muscle strength will be measured using hand-held dynamometry (Maximal voluntary force during knee extension).
Modified Sit-to-Stand Test (between-group change) | RCT: Pre-intervention (6-18 months post-stroke) and post-intervention (12-24 months post-stroke).
  This test is a modified version of the classic 5-times chair rise test. Participants will perform 5 sit-to-stand movements as fast as possible but will be provided with body weight unloading to facilitate a more appropriate movement intensity allowing them to finish within 60 second. Thus, this is a performance-based measurement.
Blood Biomarkers (between-group change) | Cohorte: 3 months post-stroke. RCT: Pre-intervention (6-18 months post-stroke) and post-intervention (12-24 months post-stroke).
  Blood samples will be drawn 3 months post stroke and pre- and post-intervention (6 and 12 months post-stroke). Samples will be analysed using single-molecule arrays (simoa) to determine blood concentrations of neurofilament light chain and glial fibrillary acidic protein and changes in peripheral blood mononuclear cells using flow cytometry
Modified Ashworth Scale (between-group change). | RCT: Pre-intervention (6-18 months post-stroke) and post-intervention (12-24 months post-stroke).
  The Modified Ashworth Scale is clinical assessment of spasticity defined as velocity-dependent exaggeration of stretch reflexes. Change in muscle tone is assessed on a 6-point ordinal scale by moving the joints of the participants through full range of motion at a standardised velocity with ratings ranging from 0 (no increase in tone) to 4 (limb rigid in flexion and extension)
Oxford Cognitive Screen (between-group change) | RCT: Pre-intervention (6-18 months post-stroke) and post-intervention (12-24 months post-stroke).
  The Oxford Cognitive Screen (OCS) is a stroke-specific cognitive test with 5 domains: Attention and executive function, language, memory, number processing, and praxis. All tasks are scored individually and can be compared against normative data to determine impairments.
Montreal Cognitive Assessment (between-group change) | RCT: Pre-intervention (6-18 months post-stroke) and post-intervention (12-24 months post-stroke).
  The Montreal Cognitive Assessment (MoCA) is a dementia screening tool commonly used in clinical trials to screen for cognitive deficits following stroke. The MoCA tests the following cognitive domains and provides a total score from 0-30, where 30 indicates best possible cognitive function: visuospatial abilities, executive functions, short-term memory recall, attention, concentration, working memory, language, and orientation to time and space.
Major Depression Inventory (between-group change) | RCT: Pre-intervention (6-18 months post-stroke) and post-intervention (12-24 months post-stroke).
  The Major Depression Inventory is a dual function questionnaire (diagnostic tool or rating scale). In the present study it is used as a rating scale to indicate the degree of depression on a scale from 0 (no depression) to 50 (maximum depression).
MRI-scans | RCT: Pre-intervention (6-18 months post-stroke) and post-intervention (12-24 months post-stroke).
  Magnetic Resonance Imaging (MRI) will be used (Structural and resting-state functional MRI scans)
MoCap | RCT: Pre-intervention (6-18 months post-stroke) and post-intervention (12-24 months post-stroke).
  Motion capure will be used to perform a 3-dimensional gait analysis during the gait test and sit-to-stand test. Kinematics and temporospatials will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Jon Skovgaard Jensen, Ph.d.-student, Principal Investigator — Department of Clinical Research, University of Southern Denmark; Anders Holsgaard-Larsen, Professor, Study Director — Odense University Hospital and Department of Clinical Research, University of Southern Denmark
Locations (2):
- Denmark (2):
  - Rigshospitalet and Herlev Gentofte Hospital, Copenhagen
  - Odense University Hospital, Odense

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Skovgaard Jensen J, Sorensen AS, Kruuse C, Nielsen HH, Skov CD, Jensen HB, Buckwalter MS, Bojsen-Moller J, Lambertsen KL, Holsgaard-Larsen A. The effect of robot-assisted versus standard training on motor function following subacute rehabilitation after ischemic stroke - protocol for a randomised controlled trial nested in a prospective cohort (RoboRehab). BMC Neurol. 2024 Jul 4;24(1):233. doi: 10.1186/s12883-024-03734-9. PMID 38965499